CLINICAL TRIAL: NCT04225455
Title: The Use of the Dexcom G6® in Commercial Pilots With Insulin-treated Diabetes (DEXFLY2)
Brief Title: The Use of the Dexcom G6® in Commercial Pilots With Insulin-treated Diabetes
Acronym: DEXFLY2
Status: Active, not recruiting | Type: Observational
Sponsor: University of Surrey (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Protocol version 6.1 21OCT2022
Record Dates: First submitted 2020-01-02; First posted 2020-01-13 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Insulin Dependent Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Glucose monitoring — To compare the glucose monitoring CGMS Dexcom G6® with their usual self-glucose monitoring in pilots by way of assessing times achieved in safe Green flying range, in Amber flying range and in Red flying range as defined by the ARA.MED.330 diabetes protocol.
  [Green: 5-15 mmol/L; Amber: 4 to <5mmol/L and >15 to 20mmol/L; Red: <4mmol/L and >20mmol/L]

SUMMARY:
To compare glucose control achieved by using real time continuous glucose monitoring (CGMS) Dexcom G6® in combination with self-monitored blood glucose during flight and also with free living in pilots.

DETAILED DESCRIPTION:
People with diabetes sometimes consider that they are subjected to unfair discrimination in the occupational or work environment. These include safety-critical activities such as operating machinery and driving. Some occupations preclude the use of medications that lower blood glucose, particularly insulin. Safety regulators, occupational health physicians and national organisations frequently have to balance the competing priorities of individual rights against public safety.

Modern treatment, with advances in insulin therapy and glucose monitoring, combined with rigorous clinical assessment and review, has allowed stereotypical attitudes to be challenged, and advocated individual assessment with respect to safety criteria. Several national authorities (Australia, Canada, UK, and USA) have, over recent years, allowed private pilots to fly for recreation while receiving treatment with insulin Canada (in 2002) was the first country to allow commercial pilots, treated with insulin, to fly commercially and have granted licences to a small number of insulin-treated pilots on a case-by-case basis and subject to close supervision.

In 2010 the UK Civil Aviation Authority (CAA) convened an expert committee to review current scientific knowledge and international policies concerning flying. The committee advised that a protocol for safe flying could be developed and produced the first iteration with subsequent refinement. It was decide that continuous glucose monitoring systems (CGMS) did not provide an accurate measurement of glucose, thus, finger prick-blood glucose monitoring was thought to provide accurate blood glucose measurement and was stipulated in the protocol (4). In 2012 the UK CAA started issuing EU Class 1 medical certificates for commercial flying to pilots with insulin-treated diabetes, having published a rigorous protocol and started collecting data systematically. Ireland and Austria have subsequently joined the protocol. The protocol has been shown to be feasible, practical and to date no safety concerns have arisen. The results from the first 26 pilots have been presented at the annual EASD conference and published in The Lancet Diabetes & Endocrinology (5). A copy of the policy is attached in appendix 1 "UK CAA policy for the Medical Certification of Pilots and Air Traffic Controllers (ATCOs) with Diabetes". In summary, the policy describes that pilots have to be in good health in terms of diabetes and associated diseases of cardiovascular system.

There should be a log book of the glucose monitoring results with each pilot at all times. The protocol suggests that the logged data will be checked against the stored memory of the glucose meters from time to time to ensure accurate data collection. The Aircrew Regulation (European Commission Regulation (EU) 1178/2011) was amended in 2015 with the inclusion of ARA.MED.330 'Special Medical Circumstances' in Annex VI (Part ARA). This allowed research to be carried out to gather evidence on the safe exercise of privileges when new medical developments (eg treatment, procedures or new medical technology) are identified that may justify a fit assessment of applicants who would not otherwise comply with certificatory requirements. This amendment was not included in the Air Traffic Control Officer (ATCO) regulations. The detailed text is available in and easy access form issued by the European Aviation Safety Agency (EASA) in May 2019.

RATIONALE We believe that reliable CGMS will have significant benefits such as access immediate access to the glucose results to the pilots, which will help them reliably to decide and adjust the insulin requirements both at flying and in free living giving rise to a controlled glucose monitoring. The pilots from UK and Austria and Ireland who have been approached are universally keen to help with any initiative that may promote safety and acceptance of the ARA.MED 330 diabetes protocol.

We wish to explore the use of the Dexcom G6® in pilots with insulin-treated diabetes, who are flying commercial aircraft with Class 1 and flying instructors or private pilots with class 2 certificates.

RESEARCH QUESTION/AIM(S) We propose that the use of continuous glucose monitoring (CGM) employing a current sophisticated device will give pilots valuable additional information about the control of their diabetes that will enhance their safety while flying. Pilots state that having immediate access to information of trends in falls or elevations in blood glucose would complement the current protocol for measurement of capillary blood glucose obtained by finger prick. We surmise that pilots will be much better equipped to manage their diabetes during flight.

STUDY DESIGN and METHODS of DATA COLLECTION AND DATA ANALYSIS This will be an observational study comparing the use of the factory calibrated real-time glucose monitoring Dexcom G6® with other glucose monitoring systems, in pilots with insulin-treated diabetes, who are flying commercial aircraft with Class 1 and flying instructors or private pilots with class 2 certificates. Dexcom G6® is CE marked, CE591560. Participants (pilots) will be blinded to the continuous monitoring glucose data from Dexcom-G6® for the first month followed by further 5 months where the participants will be encouraged to use the data from CGMS Dexcom-G6® for self-glucose monitoring alongside the usual approved protocol by the CAA. The involvement of the pilots in the study will be 12 months

The purpose of blinding is to be in line with the requirements of the ARA.MED.330 amendment to the regulation. This will allow us to investigate whether or not the pilots can maintain a stable blood glucose concentration in accordance to the CAA protocol while blinded to the glucose monitoring of Dexcom G6® but wearing the sensor as in the study design condition and if their recorded data would agree with the results recorded from Dexcom G6®.

Screening visit (visit ; Day-1) All pilots due in for their usual CAA required medical assessment will receive a copy of the PIS with the usual clinic invitation by post two weeks prior to the visit. The administration staff at the CAA, Aviation House, will be provided with copies of the PIS for this study and will be asked to include a copy of the PIS in the clinic invites.

Pilots will be asked to the CAA clinic. Before screening takes place participants will be provided with verbal and written information about the trial and the procedures involved. The pilots will be fully informed of their responsibilities and rights while participating in this exploratory trial. They will be given the opportunity to ask questions and ample time to consider participation. Participants who wish to participate in the trial will be required to sign and date an Informed Consent Form prior to any trial-related activities taking place. The PI on the site will seek informed consent from the participants. All participants will be provided with a copy of the Participant Information Sheet and of their own signed and dated Informed Consent Form.

At the screening visit the following will be performed and recorded: medical history, current medication, physical examination, diastolic and systolic blood pressure, heart rate, weight, height, age, tobacco smoking status, alcohol intake, both clinical chemistry (lipid profile, creatinine, ACR), HbA1c results required for the clinic visit, previous 6 month self-monitoring glucose data. If the participant fulfils all inclusion criteria and none of the exclusion criteria they will be accepted into the study.

Visit 1: Pilots who are eligible for the study, whether or not using a continuous glucose monitoring or Flash glucose monitoring (CGMS/FGM) (potentially will be running two devices for 6 months, current and DEXCOM-G6®), following screening will have a 1:1 training session with a research fellow skilled in diabetes, on fitting the sensor under the skin and monitoring blood glucose by Dexcom-G6® device. The participants will be informed that they will be required to wear the sensor under the skin at all times during the next 180 days of the study.

All participants will be instructed to use the CGMS Dexcom-G6® alongside their usual glucose monitoring and CGMS/FGM for 1 month during which the participants will be blinded from the Dexcom-G6® results. This blinded period acts as a baseline to understand glucose levels that are being experienced by the participants prior to introduction of the monitor.

Participants will be asked to fill in the baseline Quality of Life / Patient Related Outcomes (QOL/ PRO) questionnaires: Bolus Insulin Questionnaire, Care Management Time Form, CGM Attitudes, CGM Expectations Questionnaire, CGM Satisfaction Scale, Clarke Hypoglycaemia Awareness Survey, Diabetes Distress Scale (DDS), Diabetes Numeracy Test (DNT5), Health Questionnaire (EuroQol Group), Health Service Utilization Form, Hypoglycaemic Fear Survey, Worry subscale (HFS-W), Hypoglycaemia Confidence Scale, WHO-5 Well-Being Index, WHO-5 Well-Being Index. The questionnaires are validated and proven to be useful to evaluate CGM in other studies in subjects with diabetes.

Visit 2: This telephone call visit will take place after 6 month (Day- 180±7). Participants will be contacted by telephone with prior appointment, made on visit 1. At this Tele- visit, the participants will be asked on how they managed the fitting and wearing the rtCGMS Dexcom 6 ® and if they were happy to carry on with the study. They will then be unblinded to the rtCGMS. The participants will be allowed to use the Dexcom G6® glucose monitoring data and may choose to discontinue using other forms of CGMS/FGM if they wish. They will be encouraged to use the CGMS Dexcom G6® as much as possible to achieve good glucose control and limit episodes of hyper and hypoglycaemia, both while free living and while flying. Finger-prick glucose monitoring will carry on during the study alongside the use of the Dexcom G6® and will be logged in the pilots' log book as per CAA protocol. The data from the Dexcom-G6® will be reviewed in the next usual clinic visit.

Visit 3: This will take place at the end of 12 months (Day- 360±7).

Pilots will be asked to attend their usual clinic appointment The following will be reviewed and measured: medical history, current medication, physical examination, diastolic and systolic blood pressure, heart rate, weight, alcohol intake, clinical chemistry (lipid profile, creatinine, ACR), HbA1c required for the clinic visit. The data from the CGMS Dexcom-G6® will be reviewed and collected. The capillary glucose monitoring data recorded in the participants' log books will also be collected. We will also collect the data generated from the other CGMS devices that the participants wished to carry on using alongside Dexcom G6®.

Participants will be asked to fill in the Quality of Life / Patient related outcomes (QOL/ PRO) questionnaires at the end of the study.

Measurements:

Visits 1&3 Participant's height will be taken on Visit 1 and weight will be measured on each occasion. Vital signs, blood pressure, heart rate will also be measured on Visit 1 and Visit 3.

Recordings:

Visits 1 and 3 Laboratory investigation are carried out by local hospital laboratories according to the CAA protocol.

The results of the glucose, lipid profiles, creatinine concentrations, albumin to creatinine ratio (ACR) and HbA1c, required for the usual CAA clinic visit will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 y inclusive.
* Any ethnicity
* Pilots requiring insulin replacement therapy
* Pilots holding a class 1 or class 2 certificate
* Pilots currently participating in the current scheme
* Able and willing to perform self-blood glucose monitoring.
* Able and willing to wear a Continuous Glucose Monitoring System (CGMS) for 6months

Exclusion Criteria:

* Outside of stated age range.
* Those who are part of the protocol but are not flying currently.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 pilots with class 1 and flying instructors or private pilots with class 2 medical certificates with insulin dependent diabetes
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
To compare the data generated from the continuous glucose monitoring system (CGMS) Dexcom G6® with their routine self-glucose monitoring in pilots with class 1 and class 2 certificates | At the end of 6 months monitoring of each pilot. There will be an interim data analysis with the data collected from 25 pilots and the main analysis will be conducted once all participants have completed monitoring period within 12 months
  At visit 1 at the Civil Aviation Authority (CAA)- CGMS Dexcom G6® measures capillary glucose concentration continuously via a sensor secured under the skin. The glucose concentration is then transmitted to a hand held receiver and uploaded regularly, these data will be used to monitor glucose concentration at all times by the pilots except for the blinded period. The pilots will be blinded to the receiver data during the first month of the trial but will be unblinded there on so they will be able to see the glucose readings on the receiver for the next 5 months. The data generated from the CGMS Dexcom G6® will be compared with the routine self-glucose monitoring recorded in the log books in pilots by way of assessing times achieved in safe Green flying range, in Amber flying range and in Red flying range as defined by the ARA.MED.330 diabetes protocol.
  [Green: 5-15 mmol/L; Amber: 4 to <5mmol/L and >15 to 20mmol/L; Red: <4mmol/L and >20mmol/L]

SECONDARY OUTCOMES:
Glucose variability while flying | At the end of 6 months monitoring of each pilot. There will be an interim data analysis with the data collected from 25 pilots and the main analysis will be conducted once all participants have completed monitoring period within 12 months
  The pilots will be asked to mark the flying time as an event on the receiver while on the 6-month trial with CGMS Dexcom G6. This will allow us to compare the glucose monitoring CGMS Dexcom G6® with their routine self-glucose monitoring while flying during the blinded or unblinded period by way of assessing times achieved in safe Green flying range, in Amber flying range and in Red flying range as defined by the ARA.MED.330 diabetes protocol.
  [Green: 5-15 mmol/L; Amber: 4 to <5mmol/L and >15 to 20mmol/L; Red: <4mmol/L and >20mmol/L]
Glucose variability during non-flying normal living | At the end of 6 months monitoring of each pilot. There will be an interim data analysis with the data collected from 25 pilots and the main analysis will be conducted once all participants have completed monitoring period within 12 months
  As flying times are marked on the receiver we will also be able to compare the glucose monitoring CGMS Dexcom G6® data during the non-flying normal living with the routine self-glucose monitoring during the blinded or unblinded period by way of assessing times achieved in safe Green flying range, in Amber flying range and in Red flying range as defined by the ARA.MED.330 diabetes protocol.
  [Green: 5-15 mmol/L; Amber: 4 to <5mmol/L and >15 to 20mmol/L; Red: <4mmol/L and >20mmol/L]
Clinical chemistry data- HbA1c | At the end of 6 months monitoring of each pilot. There will be an interim data analysis with the data collected from 25 pilots and the main analysis will be conducted once all participants have completed monitoring period within 12 months
  At visit 1 and visit 3, which occurred at the standard CAA required 6 month clinic visit of the pilots, point-of-care HbA1c test results will be recorded from the clinic notes at the CAA. The data collected from the baseline will be compared with the data collected at 6 months.
Previous 6 months logged data | At the end of 6 months monitoring of each pilot. There will be an interim data analysis with the data collected from 25 pilots and the main analysis will be conducted once all participants have completed monitoring period within 12 months
  At visit 1, the previous 6 months figure-stick self-glucose monitoring data from the pilots' log books will be recorded. The previous 6 months data will be compared with the data collected with CGMS Dexcom G6 and the accompanied fingerstick glucose measurements from the pilots' log books.

CONTACTS AND LOCATIONS:
Overall Officials: David Russell-Jones, MD PhD, Principal Investigator — University of Surrey
Locations (1):
- University of Surrey FHMS Nutritional Sciences, Guildford, Surrey, United Kingdom

REFERENCES:
- [Background] Garden GL, Shojaee-Moradie F, Hutchison EJ, Frier BM, Shaw KM, Heller SR, Koehler G, Mader JK, Maher D, Roberts GA, Russell-Jones DL. Continuous Glucose Monitoring by Insulin-Treated Pilots Flying Commercial Aircraft Within the ARA.MED.330 Diabetes Protocol: A Preliminary Feasibility Study. Diabetes Technol Ther. 2023 Aug;25(8):543-548. doi: 10.1089/dia.2023.0069. PMID 37384853
- [Background] Garden GL, Fan KS, Paterson M, Shojaee-Moradie F, Borg Inguanez M, Manoli A, Edwards V, Lee V, Frier BM, Hutchison EJ, Maher D, Mathieu C, Mitchell SJ, Heller SR, Roberts GA, Shaw KM, Koehler G, Mader JK, King BR, Russell-Jones DL; EASA Diabetes Consortium. Effects of atmospheric pressure change during flight on insulin pump delivery and glycaemic control of pilots with insulin-treated diabetes: an in vitro simulation and a retrospective observational real-world study. Diabetologia. 2025 Jan;68(1):52-68. doi: 10.1007/s00125-024-06295-1. Epub 2024 Nov 4. PMID 39496965